CLINICAL TRIAL: NCT05316077
Title: Safety and Performance of Vectorio® in Conventional Trans-Arterial Chemo-Embolization (cTACE): A Post-Market Clinical Follow-up
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Other Study IDs: VEC-88-001
Record Dates: First submitted 2022-03-18; First posted 2022-04-07 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vectorio® kit

SUMMARY:
This study is conducted within the frame of the Post-Market Surveillance (PMS) activities, as described in the Post Market Clinical Follow-up (PMCF) plan of Vectorio®. This study aims at collecting clinical data, to confirm the General Safety and Performance Requirements of Vectorio® which is a Lipiodol Resistant Mixing & Injection System for cTACE.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male adult patient older than 18 years
2. Patient with confirmed diagnosis of HCC and eligible for cTACE procedure
3. Patient affiliated to national health insurance according to local regulatory requirements
4. Patient having read the information and having provided his/her consent to participate in writing by dating and signing the informed consent form

Exclusion Criteria:

1. Patient with contraindications to cTACE procedure
2. Patient with known contra-indication(s) to the use or with known sensitivity to Lipiodol or chemotherapeutic agent
3. Pregnant or breast-feeding female patient.
4. Patient unlikely to comply with the CIP, e.g. uncooperative attitude and unlikelihood of completing the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with confirmed diagnosis of hepatocellular carcinoma (HCC) and eligible for cTACE procedures
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Rate of leakage/breakage | During cTACE procedure

SECONDARY OUTCOMES:
Time necessary to obtain a water in oil emulsion defined as time between the filling of 20 mL-syringe with Lipiodol (T0) and the obtention of water in oil emulsion ready for injection (Te). | During cTACE procedure
  Collection of the time needed to obtain water in oil emulsion (Lipiodol/chemotherapeutic agent)
Ease of emulsion preparation through a rating scale | During cTACE procedure
  Rating scale: 0: Difficult - 1: Easy - 2: Very Easy (if rating is difficult, reason should be specified)
Need to perform remixing during cTACE procedure | During cTACE procedure
  Need to perform remixing : Yes/No - If Yes, how many times: Once, twice, three times, more
Assessment of per procedure Lipiodol tumor uptake rate by angiography and/or Cone Beam CT | During cTACE procedure
  Lipiodol tumor uptake: 0-25%; 25-50%; 50-75%; 75-100%
Collection of Adverse Device Effects (ADEs)/Serious Adverse Device Effects (SADEs) /Device Deficiencies (DDs) | Study period

CONTACTS AND LOCATIONS:
Locations (3):
- Univ.-Klinik für Radiologie, Graz, Austria
- CHU-Hôpital François Mitterrand, Dijon, France
- CHUV, Lausanne, Switzerland